CLINICAL TRIAL: NCT00922389
Title: A Randomized, Controlled, Parallel Design, Safety and Efficacy Study of Granulocyte Colony Stimulating Factor Mobilized Autologous Peripheral Blood Mononuclear Cell Therapy in Subjects With Diabetic Limb Ischemia.
Brief Title: A Clinical Trial on Diabetic Foot Using Peripheral Blood Derived Stem Cells for Treating Critical Limb Ischemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beike Biotech India Pvt.ltd (Industry)
Responsible Party: Director, Beike Biotech India Pvt.ltd
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNS-P0-V1
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2009-06-17 (Estimated); Status verified 2009-06

CONDITIONS: Diabetic Foot; Critical Limb Ischemia; Leg Ulcers
Keywords: Diabetes Complications; Lower limb ischemia; Adult stem cells; peripheral blood stem cells
MeSH Terms: conditions — Diabetic Foot; Chronic Limb-Threatening Ischemia; Leg Ulcer; Diabetes Complications | interventions — Granulocyte Colony-Stimulating Factor; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- G-CSF + Stem cells (Experimental)
  Interventions: Procedure: will receive G-CSF and peripheral blood derived mononuclear cells
- No stem cell group (Other)
  Interventions: Drug: G-CSF
- Standerd theraphy (Active Comparator): Any therapy for diabetic foot CLI which is routinely practiced and accepted in India
  Interventions: Drug: Standard Therapy

INTERVENTIONS:
Procedure: will receive G-CSF and peripheral blood derived mononuclear cells — Multiple intra muscular implantation of mononuclear stem cells derived from peripheral blood after G-CSF (granulocyte colony-stimulating factor)mobilization in either of two individual dose ranges which would be given to equal number of subjects.
  Arms: G-CSF + Stem cells
Drug: G-CSF — 5 micrograms/kg/day for 4 days by subcutaneous route
  Arms: No stem cell group
Drug: Standard Therapy — Any thing directed to improve blood perfusion in the limb example.Heparin,Antiplatelet agents etc
  Arms: Standerd theraphy

SUMMARY:
The purpose of this study is to determine whether the method (implanting stem cells derived from peripheral blood after G-CSF mobilization) of treatment is safe and effective in the management of diabetic foot ischemia, the therapeutic effect of stem cells is caused by improving blood circulation in ischemic limb which would in turn promote ulcer healing, prevent amputation of limb and relieve the Sevier pain of ischemia.

DETAILED DESCRIPTION:
One devastating complication of diabetes is peripheral arterial disease (PAD) including critical limb ischemia (CLI), which may result in limb loss. Epidemiological evidence confirms an association between diabetes and increased prevalence of peripheral arterial disease (PAD). The prevalence of peripheral vascular disease among the Indian diabetic population is 13%.

This therapy provides a targeted approach i.e. by improving blood perfusion in the ischemic area of the lower limb by inducing neovascularization, which would be further evaluated by measuring the change in transcutaneous partial pressure of oxygen (TCpO2), NMR angiography of local vessels, ulcer healing, pain relief, limb salvage, ABI index etc.

The specific design of the trial enables us to differentially study the effect of stem cell on diabetic foot CLI as compared to G-CSF (granulocyte colony stimulating factor) in (one control group) and standard therapy (in another control group), this study would also evaluate the effect of stem cell dose.

Extracting stem cells from this method is far more easy to perform as compared to extracting from bone marrow and is less painful for the patient as well.

The yield of mononuclear stem cell from peripheral blood is much higher as compared to bone marrow and role of CD34+ cells in limb ischemia is not yet established in humans, therefore this study would evaluate the dynamics of different types of mononuclear cells and its correlation with the therapeutic effect.

This clinical trial highlights the safety of using G-CSF in diabetic CLI by having a separate control group in which volunteers would be given only G-CSF through subcutaneous route, also this would tell about the therapeutic effect if any attributable to it.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic patients with controlled blood sugar levels
* Subject has an Ankle-brachial index < 0.6
* TCpO2 < 30-45 mm Hg measured at the calf muscle
* Subjects with unilateral or bilateral diabetic critical limb ischemia (reduced TCpO2 (<30-45 mm Hg)) who are:

  * Non reconstructable PAD as assessed by a qualified vascular surgeon on case to case basis depending upon results of angiography and clinical judgment.
  * Subjects not likely to be benefited with prostaglandin E1
* Lower extremity Ulcers of Grade II of Wagner's classification
* All subjects test negative for human immunodeficiency virus, hepatitis B virus, hepatitis C virus and treponema pallidum and their respective antibodies
* S Creatinine < 2.5 mg/dL
* All female participants in the study should be practicing a medically acceptable form of contraception (IUD, the pill etc.)
* Subject has had previous conservative treatment which resulted in little or no improvement
* Subject has had no stem cell treatment within the past 6 months o Subject is competent to provide informed consent and follow study procedures and instructions

Exclusion Criteria:

* All the subject below age 18 years and above 65 years.
* The presence of Ischemic ulcers with infectious symptoms anywhere on the lower extremity (Grade 3 and above of Wagner classification would be excluded from the study in the screening period)
* Diabetes mellitis with HbA1c > 8.5% or associated with proliferative retinopathy
* Any past or present malignancy
* Susceptibility to severe allergic reactions or a history of severe allergic reactions
* Recent occurrence (within 3 months) of myocardial infarction or brain infarction
* Coronary angioplasty within the past 1 year
* Atrial fibrillation or presence of mechanical mitral prosthetic valve
* Presence of uncontrolled systemic infection or its ongoing treatment
* Existing vital organ dysfunctions, including heart, lung or kidneys
* Coagulation disorders such as hemophilia, etc
* Use of any medication relevant to revascularization or perfusion
* Lactating female with a breastfeeding child
* A positive pregnancy test in female subjects
* A presence of any other significant medical risk or a suspicion of future non-compliance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-07; Primary Completion 2010-01 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Adverse events and laboratory parameters | 12 Months after the theraphy

SECONDARY OUTCOMES:
Trans Cutaneous partial pressure of Oxygen: TCpO2 | 12 Months post thraphy

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Anoop Misra, MD, Principal Investigator — Fortis FLT.LT.Rajan Dhall Hospital ,New Delhi, India; Dr.DAI ., Study Director — Beike Biotech
Locations (1):
- Fortis FLT.LT.Rajan Dhall Hospital, New Delhi, National Capital Territory of Delhi, India